CLINICAL TRIAL: NCT02655887
Title: The BARD® VENOVO™ Venous Stent Study - A Prospective, Non-Randomized, Multi-Center, Single-Arm Study of the Treatment of Iliofemoral Occlusive Disease - an Assessment for Effectiveness and Safety (VERNACULAR)
Brief Title: BARD® The VENOVO™ Venous Stent Study for Treatment of Iliofemoral Occlusive Disease
Acronym: VERNACULAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-14-007
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: May-Thurner Syndrome; Peripheral Vascular Disease; Venous Disease; Iliofemoral Occlusive Disease
Keywords: Vernacular; Iliofemoral Occlusive Disease
MeSH Terms: conditions — May-Thurner Syndrome; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- VENOVO™ Venous Stent. (Experimental): Implant of the VENOVO™ Venous Stent
  Interventions: Device: VENOVO™ Venous Stent

INTERVENTIONS:
Device: VENOVO™ Venous Stent — VENOVO™ Venous stent placement

SUMMARY:
The BARD® Venovo™ Venous Stent Study is a non-randomized clinical study intended to collect confirmatory evidence of the safety and effectiveness of the Venous Stent for the treatment of iliofemoral occlusive disease.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, single-arm clinical study of the VENOVO ™ Venous Stent for the treatment of iliofemoral occlusive disease. The study will be conducted at a maximum of 35 investigational sites ("sites") in the United States, and Europe and Australia/New Zealand. Enrollment will continue until a maximum of one hundred seventy (170) subjects are treated with the VENOVO™ Venous Stent, which is an estimated three-hundred forty (340) consecutive subjects in a non-randomized fashion. It is assumed that approximately 50% of the treated subjects will be U.S. subjects. Clinical follow-up for all treated subjects will be performed at hospital discharge, 30-days, and 6-, 12-, 24-, and 36-months post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The subject provides written informed consent using an Informed Consent Form approved by Ethics Committee/ Institutional Review Board for the site.
2. Subject agrees to comply with the protocol-mandated follow-up procedures and visits.
3. The subject is a male or non-pregnant female ≥ 18 years old with an expected lifespan sufficient to allow for completion of all study procedures.
4. The subject has symptomatic (non-malignant) venous outflow obstruction in iliofemoral "venous segments".
5. The subject has symptomatic venous outflow obstruction (non-malignant) in iliofemoral venous segments(Clinical-Etiology-Anatomic-Pathophysiologic (CEAP) "C" ≥ 3 or VCSS pain score of ≥ 2).
6. The subject is able and willing to comply with any required medication regimen.
7. The reference vessel diameters are between 7mm and 19 mm.

Exclusion Criteria:

1. Subject is unable or unwilling to provide written informed consent, or is unable or unwilling to conform to the study protocol follow-up procedures and visits.
2. Subject is or plans to become pregnant during the study.
3. Subject has contralateral disease of the common femoral vein, external iliac vein, common iliac vein, or any combination thereof and does not meet the venous outflow obstruction requirement or has a malignant obstruction.
4. The subject is asymptomatic, has a CEAP "C" <3, or a VCSS pain score of <2.
5. The subject has a venous obstruction that extends into the inferior vena cava (IVC) or below the level of the lesser trochanter.
6. The subject has a known uncorrectable bleeding diathesis or active coagulopathy.
7. The subject has a known allergy or sensitivity to Nickel or Titanium or intolerance to antiplatelet, anticoagulant or thrombolytic medications medications required per the protocol
8. The subject has a known allergy or sensitivity to contrast media, which cannot be adequately pre-medicated.
9. The subject has any planned surgical interventions within 30 days prior to, or within 30 days after the planned study procedure.
10. The subject has a lesion or occlusion which cannot be traversed with a guidewire.
11. The subject has had prior stenting in the target vessel.
12. The subject has iliofemoral venous segments unsuitable for treatment with available sizes of study devices.
13. The subject has another medical condition, which may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow completion of study procedures and follow ups.
14. The subject is currently participating in an investigational drug, biologic, or another device study.
15. The subject is currently on dialysis or has a serum creatinine ≥2.5mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dake, MD, Principal Investigator — Lead Principal Investigator
Locations (21):
- United States (12):
  - Vascular Breakthroughs, LLC, Darien, Connecticut
  - Yale University, New Haven, Connecticut
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Metro Health Hospital, Wyoming, Michigan
  - Cox Medical Centers, Springfield, Missouri
  - Mount Sinai Medical Center, New York, New York
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Centra Health, Inc., dba Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Sentara Medical Group, Virginia Beach, Virginia
  - Lake Washington Vascular, PLLC, Bellevue, Washington
  - CAMC Health Education and Research Institute, Charleston, West Virginia
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - JMLS Medical Services PTY LTDT/A PERTH INST. of VASCULAR RESEARCH, Perth, Western Australia
- Germany (3):
  - Uniklinik RWTH, Aachen
  - Klinikum Arnberg, Arnsberg
  - Universitaets-Herrzentrum Freiburg-Bad Krozingen, Bad Krozingen
- University Hospital Galway, Galway, Ireland
- MUMC Maastricht, Maastricht, Netherlands
- Fundacion de investigacion HM Hospitales, Madrid, Spain
- Guy's & St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Dake MD, O'Sullivan G, Shammas NW, Lichtenberg M, Mwipatayi BP, Settlage RA; VERNACULAR Trial Investigators. Three-Year Results from the Venovo Venous Stent Study for the Treatment of Iliac and Femoral Vein Obstruction. Cardiovasc Intervent Radiol. 2021 Dec;44(12):1918-1929. doi: 10.1007/s00270-021-02975-2. Epub 2021 Sep 20. PMID 34545448

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated at 25 investigational sites in the U.S., Europe and Australia. First subject was enrolled June 15, 2016, and the last subject on May 1, 2017. Approximately 60% of subjects are in the U.S.
Pre-assignment Details: Three U.S. sites were activated, but did not consent subjects. A fourth site enrolled 1 subject who was lost to follow-up after discharge (site closed). Fifty-eight (58) screen failures reported and three (3) eligible subjects were not treated with the device. In total, 170 subjects were treated with VENOVO.
Period: Overall Study
Arm/Group | VENOVO™ Venous Stent.
Started | 170 (Intent to Treat (ITT) population.)
Completed | 156 (Completed 12-month follow-up.)
Not Completed | 14
Not completed — Lost to Follow-up | 3
Not completed — Death | 4
Not completed — Withdrawal by Subject | 3
Not completed — Missed 12-month follow-up visit | 4

BASELINE CHARACTERISTICS:
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 125
  ≥ 65 years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 158
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 156
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 8
  United States | 100
  Ireland | 4
  United Kingdom | 8
  Australia | 5
  Germany | 34
  Spain | 11
Cardiovascular Disease [Count of Participants; unit: Participants] — Intent to Treat (ITT) Population
  Participants
    Stroke | 4
    Angina | 5
    Hypertension | 55
    Coronary Artery Disease (CAD) | 15
    Myocardial Infarction (MI) | 6
    Transient Ischemic Attack (TIA) | 3
    Cardiomyopathy | 3
    Vascular Heart Disease | 2
    Deep Vein Thrombosis (DVT) | 92
    May-Thurner Syndrome | 102
    Venous Valve Disease | 12
    Varicosis | 133
    Dyslipidemia | 47
    Peripheral Arterial Disease (PAD) | 18
    Atrial Fibrillation (A-FIB) | 6
    Arrhythmia (other than A-FIB) | 8
Renal Disease [Count of Participants; unit: Participants]
  Chronic Kidney Disease | 4
  Acute Renal Insufficiency | 1
  Uremia | 1
Disease Category [Count of Participants; unit: Participants]
  Post-Thrombotic Syndrome (PTS) | 93
  Non-Thrombotic Iliac Vein Lesions (NIVL) | 77
Number of Target Lesions [Count of Participants; unit: Participants]
  1 | 154
  2 | 16
Number of Study Devices Used [Count of Participants; unit: Participants]
  1 Study Device | 122
  2 Study Devices | 47
  3 Study Devices | 1
Target Limb [Count of Participants; unit: Participants]
  Right Leg | 28
  Left Leg | 142

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Patency of the Venous Stent at 12 Months Post-Index Procedure
Description: Primary patency rate at 12 months post-index procedure evaluated against a literature-derived Performance Goal (PG) of 74%. Primary patency defined as: freedom from Target Vessel Revascularization (TVR); freedom from thrombus occlusion and stenosis > 50% as measured by Duplex Ultrasound (DUS).
  Please note that both the primary effectiveness and the primary safety endpoint are considered co-primary endpoints. That is, both endpoints need to be significant to claim the study as successful.
Time Frame: 12 months post-index procedure
Population: ITT subjects. 25 subjects were excluded from the denominator due to discontinuation or other reasons prior to 12 month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 145
Participants | 128
Statistical Analysis 1: Comparison: VENOVO™ Venous Stent; Hypothesis: H0 :Primary patency rate at 12 months post-index procedure from the overall VENOVO Venous Stent (BVS) patients (PTS and NIVL combined) is at most as good as that of the PG. Ha: Primary patency rate at 12 months post-index procedure from the overall VENOVO Venous Stent (BVS) patients (PTS and NIVL combined) is better than that of PG; Test type: Non-Inferiority — PG of 74%, which was set at 10% (non-inferiority margin) below the weighted mean of primary patency (PP2) rate at 12 month at a combination of 55% (PTS) subjects at primary patency rate of 77.1% and 45% (NIVL) subjects at primary patency rate of 93.4%. When taking into consideration both co-primary efficacy and safety endpoints, with 138 BVS subjects, the overall study power is at least 85%*99%=84%; p = 0.0001, Weighted Z-statistics; Weighted Z-statistics = 88.3, 90% CI 1-sided [lower limit 82.4]

2. Primary Outcome: Number of Participants With Freedom From Major Adverse Events (MAEs)
Description: Freedom from major adverse events (MAEs) defined as: Target Vessel Revascularization; Device and/or procedure related death; Major amputation of target limb; Pulmonary Embolism which is clinically important; Vascular injury requiring surgical/endovascular intervention; Embolization /migration of stent; Device or procedure related acute DVT involving the treated limb.
  Please note that both the primary effectiveness and the primary safety endpoint are considered co-primary endpoints. That is, both endpoints need to be significant to claim the study as successful.
Time Frame: 30 days post-index procedure
Population: ITT subjects. Results adjudicated by CEC. MAEs that occurred prior to day 30 of each subject's follow-up were counted as failures toward primary safety (n= 11). Those subjects were considered not evaluable and not included in the denominator for the primary safety endpoint (total evaluable = 170 subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Participants | 159
Statistical Analysis 1: Comparison: VENOVO™ Venous Stent; Hypothesis: H0: The primary safety endpoint absence from event rate in the VENOVO Venous Stent (BVS) through 30 day at most as large as that of the PG. Ha: The primary safety endpoint absence from event rate in the VENOVO Venous Stent (BVS) through 30 day is better than that of the PG; Test type: Non-Inferiority — The primary safety endpoint was evaluated against the PG of 89% which was set at 10% (non-inferiority margin) below the literature-derived average freedom from MAE rate at 30 day of 99%. A one-side p-value is derived based on an exact binomial test. When taking into consideration both co-primary efficacy and safety endpoints, with 138 BVS subjects, the overall study power is at least 85%*99%=84%; p = 0.0322, Exact binomial test; Exact binomial test = 93.5, 90% CI 1-sided [lower limit 89.5]

3. Secondary Outcome: Endpoint With Hypothesis Testing: Index of Venous Clinical Severity Score (VCSS) From Baseline to 12 Months
Description: The Venous Clinical Severity Score (VCSS) system includes 10 clinical descriptions (pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, number of active ulcers, duration of active ulceration, size of active ulceration. and level of compliance with medical compression therapy), scored from 0 to 3 (total possible score, 30) with 0 means absent, 1 means mild, 2 means moderate and 3 means severe. Total VCSS is the sum of all VCSS assessment scores from categories for a given time point. Twelve-month data is the change between baseline score and 12-month follow-up score. Results calculated for Intent-to-Treat (ITT) subjects. Lower values represent a better outcome, that is, a level of pain less than that experienced at baseline.
Time Frame: Evaluation at 12 months post-index procedure
Population: Evaluable ITT subjects are included in this analysis.(n) varies in relation to the number of evaluable subjects. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 155
Scores on a scale | -1.7 [-1.81 to -1.49]
Statistical Analysis 1: Comparison: VENOVO™ Venous Stent; H0: The distribution at the 12-month follow-up remains unimproved compared to baseline. Ha: The distribution shifts toward lower (less pain) classes; Test type: Other; p = 0.001, t-test, 2 sided — this p value is < 0.001

4. Secondary Outcome: Endpoint With Hypothesis Testing: Index of Quality of Life (QoL) From Baseline to 12 Months
Description: The Quality of Life (QoL) assessment of Chronic Venous Insufficiency Questionnaire (CIVIC-20) is a 20-item questionnaire which provides a global index and an outline of 4 QoL dimensions - pain (4 items), physical (4 items), psychological (9 items) and social (4 items). Items are scored on a scale from 1 to 5. A low score corresponds to greater patient comfort. Total CIVIQ-20 score is the sum of all 20-item scores The score of each dimension was obtained by adding up the scores of each constituent item within that dimension. Twelve-month data is the change between baseline score and 12-month follow-up score. Results calculated for evaluable ITT subjects. Lower values represent a better outcome, that is, a better QoL than that experienced at baseline.
Time Frame: Evaluation at 12 months post-index procedure
Population: Evaluable ITT subjects were included in this analysis. (n) varies in relation to the number of evaluable subjects. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 153
Scores on a scale | -15.7 [-18.41 to -12.96]
Statistical Analysis 1: Comparison: VENOVO™ Venous Stent; Test type: Other; p = 0.001, t-test, 2 sided — p value is < 0.001

5. Secondary Outcome: Endpoint Without Hypothesis Testing: Index of CEAP at 30 Days, 6 Months, and 12 Months Post Procedure
Description: Clinical-Etiologic-Anatomic-Pathophysiologic (CEAP) Classification is a system that describes a doctor's physical exam findings for vein problem(s), the cause of the problem(s), the location in the leg, and the mechanism responsible for the manifestation of the vein problem. For Clinical classification, the clinical components indicates disease severity, ranging from none (0 points) to active ulcers (6 points).For each category of Etiology, Anatomy, and Pathophysiology classifications, at each time point, frequency of each category is reported. Subsequent clinical study reports will present CEAP at 24 and 36-months follow-up. Changes from baseline measures to given time points are presented. Lower mean scores represent an improvement from baseline measure.
Time Frame: Evaluation through 30 day, 6 months and 12 months post index procedure
Population: Evaluable ITT subjects are included in this analysis. (n) varies in relation to the number of evaluable subjects at 30 days, 6 months and 12 months. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Scores on a scale
  30 day post procedure: number analyzed (Participants) | 166
  30 day post procedure | -1.1 (1.26)
  6 months post procedure: number analyzed (Participants) | 160
  6 months post procedure | -1.3 (1.34)
  12 months post procedure: number analyzed (Participants) | 155
  12 months post procedure | -1.5 (1.33)

6. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Acute Technical Success
Description: Acute technical success is defined as successful deployment of stent(s) to intended target with adequate lesion coverage as assessed by the Investigator.
Time Frame: At time of Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Participants | 170

7. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Acute Procedure Success (ITT Subjects)
Description: Technical success is defined as no major adverse events experienced between index procedure and discharge
Time Frame: Less than 30 days post index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Participants | 168

8. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Lesion Success (ITT Subjects)
Description: Lesion Success is defined as the attainment of less or equal to 50% residual stenosis at the conclusion of the index procedure.
Time Frame: At the conclusion of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Participants | 170

9. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Freedom From Target Lesion Revascularization (TLR) (ITT Subjects)
Description: Freedom from Target Lesion Revascularization (TLR) through 30 days is specific to the first revascularization procedure of the target lesion.
Time Frame: Evaluation throrugh 30 day, 6 months and 12 months post index procedure
Population: (n) varies in relation to the number of evaluable subjects at 30 days, 6 months and 12 months. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section.
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Participants
  30 day post procedure | 164
  6 months post procedure | 161
  12 months post procedure: number analyzed (Participants) | 163
  12 months post procedure | 151

10. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Freedom From Target Vessel Revascularization (TVR) (ITT Subjects)
Description: Freedom from Target Vessel Revascularization (TVR) is defined as the first revascularization procedure of the target vessel, as determined by an Independent Core Lab. Freedom from Target Lesion Revascularization (TLR) and Freedom from TVR results are the same through the 12 month analysis as all TLRs were also TVRs in this case.
Time Frame: Evaluation through 30 days, 6 months and 12 months post index procedure
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 170
Participants
  30 days post procedure | 164
  6 months post procedure | 161
  12 months post procedure: number analyzed (Participants) | 163
  12 months post procedure | 151

11. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants Without Device Stent Fracture at 12 Months Follow-Up
Description: Stents were evaluated at the 12 month follow-up for fracture analysis. Evaluable ITT subjects are included in this analysis.
Time Frame: Evaluation at 12 months post-index procedure
Population: Evaluable ITT subjects are included in this analysis. (n) varies in relation to the number of evaluable subjects. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section.
Measure: Count of Participants; unit: Participants
Arm/Group | VENOVO™ Venous Stent.
Number analyzed (Participants) | 137
Participants
  No Device Stent Fracture at 12 months | 137
  Device Stent Fracture at 12 months | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) are presented during the 12-month follow-up period. All AEs were reviewed by the CEC and a total of 129 events were adjudicated as per the committee charter. Results for ITT subjects are reported for both SAEs and AEs. AEs that occurred through 395 days for each subject are included.
Arm/Group | VENOVO™ Venous Stent.
All-Cause Mortality (participants affected / at risk) | 4/170
Serious Adverse Events (participants affected / at risk) | 44/170
Other Adverse Events (participants affected / at risk) | 63/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VENOVO™ Venous Stent. (N=170)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Coeliac artery stenosis (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Device occlusion (General disorders) | 3 (3)
Local swelling (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 6 (6)
Vessel puncture site haematoma (General disorders) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Panic attacks (Psychiatric disorders) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Heamaturia (Renal and urinary disorders) | 1 (1)
Renal artery arteriosclerosis (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic neuropathis ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Iliac vein occlusion (Vascular disorders) | 2 (2)
Pelvic vein occlusion (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Post-thrombotic syndrome (Vascular disorders) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VENOVO™ Venous Stent. (N=170)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infraction (Cardiac disorders) | 1 (1)
Palpitation (Cardiac disorders) | 1 (1)
Endocrine ophthalmopathy (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Adverse drug reaction (General disorders) | 4 (4)
Fatigue (General disorders) | 2 (2)
Hernia (General disorders) | 1 (1)
Induration (General disorders) | 1 (1)
Injection site discoloration (General disorders) | 2 (2)
Injection site discomfort (General disorders) | 3 (3)
Injection site haematoma (General disorders) | 1 (1)
Injection site induration (General disorders) | 2 (2)
Injury associated with device (General disorders) | 1 (1)
Local swelling (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 3 (3)
Thrombosis in device (General disorders) | 4 (4)
Vessel puncture site haematoma (General disorders) | 2 (2)
Vessel puncture site haemorrhage (General disorders) | 2 (2)
Vessel puncture site pain (General disorders) | 4 (4)
Vessel puncture site swelling (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Vaginal infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 11 (11)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 4 (4)
Meralgia paraesthetica (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (4)
Sciatica (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Varicose veins pelvic (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalized (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 7 (7)
Vasospasm (Vascular disorders) | 1 (1)
Venous insufficiency (Vascular disorders) | 6 (6)
Venous stenosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to PI publication of site results, sponsor requires publication of multi-centers results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/87/NCT02655887/Prot_SAP_000.pdf